CLINICAL TRIAL: NCT01398839
Title: Safety Study of the VEGA UV-A System to Treat Ectasia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Topcon Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Organization: Topcon Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CXL-002
Record Dates: First submitted 2011-07-10; First posted 2011-07-21 (Estimated); Results first posted 2013-03-04 (Estimated); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Ectasia
MeSH Terms: conditions — Dilatation, Pathologic | interventions — Riboflavin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham Control (Sham Comparator)
  Interventions: Drug: Riboflavin
- CXL Treatment (Experimental)
  Interventions: Device: VEGA UV-A Illumination System; Drug: Riboflavin

INTERVENTIONS:
Device: VEGA UV-A Illumination System — Only subjects assigned to the treatment group will receive treatment with the UV Light
  Arms: CXL Treatment
Drug: Riboflavin — Both treatment and sham groups will receive riboflavin

SUMMARY:
The purpose of this research study is to test the safety, tolerability, and effectiveness of corneal collagen cross-linking (CXL) when used to treat ectasia.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years of age or older
* Diagnosis of Ectasia
* Presence of central or inferior steepening
* Topography consistent with ectasia
* BSCVA 20/20 or worse
* If contact lens wearer; removal of contact lenses for required period of time
* Signed informed consent
* Willingness and ability to comply with schedule for follow-up visits

Exclusion Criteria:

* Previous ocular condition that may predispose the eye for future complications or prevent the possibility of improved vision
* History of chemical injury or delayed epithelial healing
* A known sensitivity to study medications
* Nystagmus or any other condition that would prevent a steady gaze during the treatment or other diagnostic tests
* A condition that would interfere with or prolong epithelial healing
* Presence or history of any other condition or finding that makes the patient unsuitable for treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2010-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Barnet Dulaney Perkins Eye Center, Phoenix, Arizona
  - Woolfson Eye Institute, Atlanta, Georgia
  - Minnesota Eye Consultants, P.A., Bloomington, Minnesota
  - Laser and Corneal Surgery Assoc. PC, New York, New York
  - Mt. Sinai Hospital, New York, New York
  - Pamel Vision & Laser Group, New York, New York
  - Cleveland Clinic-Cole Eye Institute, Cleveland, Ohio
  - The Ohio State University College of Medicine, Columbus, Ohio
  - ReVision Advanced Laser Eye Center, Columbus, Ohio
  - Dell Laser Consultants, Austin, Texas
  - Slade & Baker Vision, Houston, Texas
  - The Eye Institute of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period started December 2010 and ended June 2012 at medical clinics throughout the country.
Pre-assignment Details: Enrolled participants were excluded from the clinical trial because they failed to meet one or more the inclusion/exclusion criteria.
Groups:
- CXL Treatment: VEGA UV-A Illumination System : Only subjects assigned to the treatment group will receive treatment with the UV Light
  Riboflavin : Both treatment and sham groups will receive riboflavin
- Sham Control: Riboflavin : Both treatment and sham groups will receive riboflavin
Period: Overall Study
Arm/Group | CXL Treatment | Sham Control
Started | 35 | 37
Completed | 35 (The study was terminated. The exact number of patients completing all visits is unknown.) | 37 (The study was terminated. The exact number of patients completing all visits is unknown.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CXL Treatment | Sham Control | Total
Number analyzed (Participants) | 35 | 37 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | NA — The study was terminated prior to data analysis. | NA — The study was terminated prior to data analysis. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Between 18 and 65 years | NA — The study was terminated prior to data analysis. | NA — The study was terminated prior to data analysis. | NA — Total not calculated because data are not available (NA) in one or more arms.
  >=65 years | NA — The study was terminated prior to data analysis. | NA — The study was terminated prior to data analysis. | NA — Total not calculated because data are not available (NA) in one or more arms.
Age, Continuous [Mean (Standard Deviation); unit: years] | NA (NA) — The study was terminated prior to data analysis. | NA (NA) — The study was terminated prior to data analysis. | NA (NA) — The sponsor terminated the study prior to data analysis for financial reasons.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — The study was terminated prior to data analysis. | NA — The study was terminated prior to data analysis. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — The study was terminated prior to data analysis. | NA — The study was terminated prior to data analysis. | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants]
  United States | 35 | 37 | 72

OUTCOME MEASURES:

1. Primary Outcome: Changes in Corneal Curvature
Time Frame: 6 Months
Population: The CXL-002 study was terminated and data analysis was not done. The sponsor, Topcon Medical Systems, decided to terminate the study for administrative reasons only, and not as a result of any safety issues or concerns relating to the study.
Arm/Group | CXL Treatment | Sham Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | CXL Treatment | Sham Control
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/37
Other Adverse Events (participants affected / at risk) | 0/35 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All such Confidential Information shall remain the property of Topcon, as applicable, and Institution agrees that neither it nor Principal Investigator nor any of its employees or Sub-Investigators, if any, shall disclose any of the Confidential Information to third parties, without the prior written consent of Topcon.